CLINICAL TRIAL: NCT07128511
Title: Compare Training Strategies to Maintain Cognitive Performance Under Respiratory Load
Brief Title: Training Strategies to Maintain Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202500759
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Shortness of Breath; Shortness of Breath/Dyspnea; Respiratory Distress
Keywords: dyspnea; shortness of breath; respiratory loading; breathing patterns
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Inhalation Breathing Pattern (Experimental): In this arm, participants use a breathing pattern consisting of brief, rapid, successive inhalations.
  Interventions: Behavioral: Multiple Inhalation Breathing Pattern
- Tactical Breathing Technique (Active Comparator): In this arm, participants use a slow, paced breathing cycle with intentional inhale-hold-exhale-hold phases.
  Interventions: Behavioral: Tactical Breathing Technique

INTERVENTIONS:
Behavioral: Multiple Inhalation Breathing Pattern — This behavioral intervention involves a breathing pattern characterized by brief, rapid successive inhalations within each breath cycle. The timing of each short inhalation is coordinated with fast, cyclical auditory tones, providing a consistent rhythm for participants to follow. Visual cues are also displayed to reinforce the timing and sequence of breaths.
  During training, participants first practice the breathing pattern without any cognitive task, followed by practice while performing the psychomotor vigilance task (PVT). The technique is then applied during the main experimental condition, where participants wear a chest wall force antagonistic device set at 25 cmH₂O to simulate the added work of breathing experienced underwater. The PVT lasts for 10 minutes, requiring participants to respond as quickly as possible to visual stimuli, allowing researchers to measure sustained attention and reaction time.
  Arms: Multiple Inhalation Breathing Pattern
Behavioral: Tactical Breathing Technique — This behavioral intervention uses a slow, paced breathing cycle incorporating four distinct phases: inhale, hold, exhale, and hold. Each phase is precisely timed and synchronized with distinct auditory tones for inhalation, hold phase, and exhalation. Participants also receive visual cues to reinforce correct timing and ensure consistency throughout the exercise.
  Training begins with participants practicing the breathing pattern without any cognitive task, followed by practice while completing the psychomotor vigilance task (PVT). The full experimental condition involves performing the 10-minute PVT while wearing a chest wall force antagonistic device set at 25 cmH₂O to simulate the restrictive breathing load experienced in underwater environments. The PVT requires quick responses to visual stimuli, allowing measurement of sustained attention and reaction time under load.
  Arms: Tactical Breathing Technique

SUMMARY:
• Statement of the Problem and Justification Cognitive performance under physiologically stressful conditions is critical in high-demand environments such as military operations, diving, and firefighting. One such stressor is restricted breathing, which can occur due to equipment (e.g., masks, regulators) or environmental pressures (e.g., underwater). Restricted breathing has been shown to increase physiological strain, which may in turn impact attention, reaction time, and task execution. Despite this, there is limited research examining how different breathing strategies can mitigate the cognitive effects of restricted respiration.

Understanding whether specific breathing techniques can preserve cognitive function under stress has practical implications for operational readiness, safety, and task performance in extreme or demanding environments.

• Synopsis of Relevant Research Previous human studies have shown that controlled breathing techniques, such as tactical or box breathing (inhale-hold-exhale-hold patterns), can reduce anxiety and improve focus in stressful situations. For example, tactical breathing has been adopted in military and law enforcement settings to enhance performance under pressure. Other research in sports psychology and respiratory therapy suggests that altering breathing frequency or depth can modulate autonomic nervous system activity, potentially affecting cognitive control and reaction time.

Additionally, psychomotor vigilance tasks (PVTs) have been widely used to assess the impact of physiological stressors - such as sleep deprivation, hypoxia, and fatigue - on sustained attention and reaction time. However, few studies have directly examined the interaction between structured breathing patterns and PVT performance during restrictive breathing loads.

• Importance and Next Step This study represents a logical next step in understanding how breathing techniques can buffer against cognitive decline under conditions that simulate real-world respiratory restriction (e.g., underwater diving). By directly comparing the effects of two distinct breathing strategies during a controlled, restrictive breathing task, this research will help determine whether certain techniques are more effective in preserving attention and reaction time. The findings could inform training and operational protocols for individuals working in challenging environments, as well as guide future studies into breathing-cognition interactions under physical stress.

DETAILED DESCRIPTION:
Study Overview This within-subject, randomized crossover study investigates how two different breathing techniques impact sustained attention during restrictive breathing conditions that simulate underwater environments. The techniques tested are a tactical combat breathing method (slow, paced breaths with intentional holds) and a multiple-breath technique involving rapid successive breaths. Each participant will perform a 10-minute psychomotor vigilance task (PVT) under each breathing pattern while in a chest wall loading device that simulates resistive breathing in underwater conditions. The order of breathing techniques will be randomized. There will be 2 visits with a rest day in between for testing two different breathing patterns.

Screening

* The general population of this experiment comprises healthy adults between the ages of 18 and 45 years.
* Subjects who consent to participate will undergo a brief screening.
* Women of childbearing age will be given a pregnancy test. If the test is positive, subjects will be excluded from the study. ·
* Study staff will fill out a demographic data sheet with the subject.
* Upright FVC (Forced Vital Capacity) will be conducted per published American Thoracic Society and European Respiratory Society (ATS/ERS) guidelines. Individuals with an FVC <75% predicted according to their age, sex, and BMI will be ineligible for further participation in this study.
* Individuals will also be excluded if they self-report any history of neurologic disease, history of cancer in the head, neck, or lungs, acute or chronic respiratory illness, use of nicotine in the past five years. When scheduling their participation, subjects will be informed to avoid eating 90 minutes before the experiment. They will also be instructed to avoid caffeine and vigorous exercise 24 hours before the experiment. Failure to do so may result in rescheduling their participation or withdrawing the subject.

Inclusion Criteria

* Age 18-45
* Healthy adult status confirmed by screening
* FVC ≥ 75% predicted (based on ATS/ERS guidelines) Exclusion Criteria
* History of neurological or respiratory disease
* Respiratory illness or recent nicotine use (within 5 years)
* Positive COVID-19 or pregnancy test Recruitment and Consent
* Participants will be recruited via flyers, email announcements, and word-of-mouth across the university campus.
* The study will include only healthy adult volunteers.
* No vulnerable populations will be targeted.
* Informed consent will be obtained by study staff in a private lab setting before participation.
* Consent will be documented and stored securely.

Study Flow and Schedule Visit 1: Orientation and Training First Pattern (Approximately 120 Minutes)

* Informed Consent and Screening Participants will review and sign an IRB-approved consent form. Forced Vital Capacity (FVC) will be assessed using a spirometer following ATS/ERS guidelines. Participants must meet the minimum criterion (≥75% predicted) to continue. Participants will also complete a brief medical and demographic questionnaire.
* Familiarization with the Chest Wall Force Antagonistic Device The device, which simulates restrictive breathing by applying external pressure to the chest and abdomen, will be introduced. In underwater diving, even when a diver breathes from a regulator supplying gas at ambient pressure, small mismatches can occur between the pressure inside the lungs and the hydrostatic pressure exerted on the chest wall. This happens when the diver tilts or changes posture, creating a vertical separation between the regulator (typically located at the mouth) and the thoracic cavity. Because hydrostatic pressure increases with depth, a vertical offset as small as 20 cm can result in a pressure difference of approximately 0.02 atm. This corresponds to about 42 pounds per square foot (psf). For a diver with a chest wall surface area of 1.6 ft², this pressure difference translates to an additional compressive force of roughly 67 pounds-force (lbf) resisting chest expansion. While subtle, such differences can increase the work of breathing and become more pronounced when restrictive gear is used or under higher respiratory loads. Understanding these effects is important for modeling respiratory mechanics and designing equipment that interacts with the chest under pressure. The subject's chest and abdominal surface area will be measured and the appropriate spring load will be used at a pressure of 25cmH20.
* Introduction ot br
* Breathing Technique Training Using Sound Cues (3 Minutes) Participants will be trained in one of two breathing techniques: 1) Tactical Breathing: Slow inhale-hold-exhale-hold cycle coordinated with auditory tones 2) Multiple-Breath Pattern: Short, successive breaths prompted by faster cyclical tones. The training is guided by both audio and visual cues to ensure timing consistency. Participants will practice first for 2 minutes with no task and then 3 minutes with the PVT task.
* Psychomotor Vigilance Task (PVT) Load Practice Trial (5 minutes x 3) Participants will complete a short (3-minute) practice version of the PVT. The task involves responding to a visual stimulus (number counter) as quickly as possible when it appears, simulating the real testing conditions. Instructions and expectations will be reviewed before beginning the experimental phase. This will also be under load conditions. There is a 2-minute recovery period between each trial. If subjects fail to follow the breathing pattern via a matching algorithm, an additional 3 minutes of training under load and an additional recovery period will be administered with a visual cue.
* Break (20 minutes)
* Psychomotor Vigilance Task (PVT) No Load Practice Trial (10 minutes) Participants will complete a 10-minute trial of the PVT task under no respiratory load while listening to the predetermined breathing pattern.
* Break (20 minutes)
* Psychomotor Vigilance Task (PVT) Load Final Trial (10 minutes) Participants will complete a 10 minute trial of the PVT task under respiratory load while listening to the predetermined breathing pattern for final trial. Physiological monitoring continues throughout. A Borg Scale will be administered after completion for questions regarding perception of task performance and load.

Visit 2: Training Second Pattern 2 Days Later (Approximately 120 Minutes)

• Same as visit 1 except for a change in breathing pattern.

Psychomotor Vigilance Task (PVT) Participants are instructed to respond as quickly as possible when a red number appears on the screen. The number represents the milliseconds elapsed since the visual cue appeared, and it stops once the participant responds. This simple, reaction-based task is widely used to assess sustained attention and is sensitive to fatigue and cognitive load.

Chest wall force antagonistic device

* In certain parts of the experiment, we will use a chest wall force antagonistic device to simulate the compression that a diver face when diving.
* This device is made of constant force springs mounted between two boards. One board is fixed, and the other moves in a sliding track. Attached to this movable board is a two-piece chest strap made of a non-flexible fabric. This fabric will go over the subject's chest wall, abdomen, and shoulders. The purpose of the movable board is to pull the chest strap with the same force that the subject would encounter if diving at 60ft underwater.
* The fabric is held together by Velcro strips. This ensures that the subject can be quickly released, if needed.
* The spring-loaded chest wall device will be set based on hydrostatic pressure difference during diving. This pressure will be 25cmH20 (or 51 lb/sf).
* If we measure the height and width of the chest wall and abdomen, we can calculate the area and the amount of pressure water would exert on their thorax and abdomen in both cases. For example, a subject with a chest wall area of 1.08sqft (12inx13in) would experience a force of 55lbs.

Interventions and Randomization

* All participants complete both breathing conditions in a randomized order.
* There is no placebo or inactive control.
* The restrictive breathing condition is created using a chest wall force antagonistic device simulating underwater load.

Physiological Measurements

* Airflow Measured using a face mask connected to a pneumotachograph and pressure transducer (Hans Rudolph). From airflow, we perform calculations for tidal volume and breathing rate during each breathing pattern.
* Mouth Pressure Collected concurrently via the same pneumotach setup to assess pressure variations during inspiration and expiration under load.
* Photoplethysmography (PPG) Infrared sensors placed on the middle fingers of both hands and ears. This provides continuous monitoring of blood volume changes and oxygen saturation (SpO2), offering real-time cardiovascular data.
* End-Tidal CO2 Measured using a line connected to the face mask. This measure provides estimates of metabolic activity and ventilation adequacy under restrictive load.
* Respiratory Inductance Plethysmography (RIP) Bands Elastic bands placed around the chest and abdomen. Used to monitor respiratory effort and expansion dynamics at both locations throughout the task. Borg Scale Questions These questions are meant to be asked about the subject's perception of load as well as cognitive performance during the experiment.
* Please rate how the pressure on your thorax is affecting your test performance.
* Please rate your level of discomfort.
* Please rate how noticeable the airway resistance is.
* Please rate how the airway resistance is affecting your test performance.
* How well do you believe you matched the breathing pattern?
* How did following the breathing pattern effect your test performance?

Comparison to Standard Therapy

* This study does not involve treatment or therapy.
* Participants may withdraw at any time without penalty.
* Participation does not impact access to any standard care or services. Statistical Analysis
* Sample Size: Target n = 15
* Primary Outcome: PVT reaction time for each subject between two breathing patterns.
* Secondary Outcome: Borg discomfort scores after each trial.
* Analyst: Data will be anonymized and analyzed by study staff. Monitoring and Oversight
* No formal DSMB required
* Safety monitored by the PI and co-investigators
* Continuous real-time monitoring of SpO2: session will be stopped if SpO2 drops below 91% or if end tidal CO2 is above 3%.
* Participants may withdraw at any time without consequence. Data Privacy and Confidentiality
* Participants will be assigned a unique ID code
* Identifiable data will be kept separate from performance data
* All electronic files will be password-protected and stored on secure servers
* Physical records will be stored in locked cabinets accessible only to approved study personnel

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Healthy adult status confirmed by screening
* FVC ≥ 75% predicted (based on ATS/ERS guidelines)

Exclusion Criteria:

* History of neurological or respiratory disease
* Respiratory illness or recent nicotine use (within 5 years)
* Positive COVID-19 or pregnancy test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task Response Time | Each trial lasts 10 minutes. There are smaller training trials for 3 minutes each.
  The Psychomotor Vigilance Task is a computer-based assessment used to measure sustained attention and reaction time. During the task, participants view a screen displaying a blank background until a visual stimulus appears. The counter represents the number of milliseconds elapsed since the stimulus appeared. Participants are instructed to respond as quickly as possible by pressing a button when the number appears, at which point the counter stops. The reaction time (in milliseconds) is recorded for each trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Malachowsky Hall for Data Science and Information Technology, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No